CLINICAL TRIAL: NCT06887127
Title: An Open-label, Long-term Extension Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of TLL-018 in Patients With Rheumatoid Arthritis
Brief Title: A Long-term Extension Clinical Study of TLL-018 in Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLL-018-304
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TLL-018 (Experimental): Participants received a two-stage treatment period in Study TLL-018-301, with treatment of 24 weeks of TLL-018 20 mg BID or tofacitinib 5 mg BID in Stage 1. In Stage 2, the participants with tofacitinib who didn't achieve ACR50 were transferred to TLL-018, and other participants maintained the original treatment. Upon completion of Study TLL-018-301, qualified participants can enter the OLE study, and all participants will receive TLL-018 20 mg BID, i.e., 2 tablets of TLL-018 10 mg orally twice daily, for 78 weeks.
  Interventions: Drug: TLL-018

INTERVENTIONS:
Drug: TLL-018 — TLL-018 20 mg BID for 78 weeks

SUMMARY:
The primary objective of the study is to evaluate the long-term safety, tolerability, and efficacy of TLL-018 in patients with rheumatoid arthritis (RA) who have completed a preceding randomized controlled trial with TLL-018.

DETAILED DESCRIPTION:
This is an open-label extension study to assess the long-term safety, tolerability, and efficacy of TLL-018 in adults with RA who have completed Study TLL-018-301(NCT06020144), a phase 3 randomized controlled trial with TLL-018.

The study includes three parts: screening period, treatment period and follow-up period. All participants will be treated with TLL-018 20 mg twice daily (BID) for 78 weeks.

Safety assessment will be conducted at 6, 12, 24, 36, 48, 60, 72, 78 weeks, including physical examination, collection of vital signs, laboratory tests, AEs, SAEs, etc.

Efficacy evaluation will be performed at weeks 12, 24, 36, 48, 60, 72, and 78, including joint assessment, PGA, PtGA, VAS, HAQ-DI questionnaires, SF-36 scale, morning stiffness assessment, DAS28-hsCRP, CDAI, SDAI, ACR20/50/70 response assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have completed TLL-018-301 study within 3 months;
* Age (at the time of consent):>＝18 years of age, <＝75 years of age;
* Female subjects of childbearing potential (WOCBP), who should not be pregnant or breastfeeding, should not enter the study until after pregnancy testing (e.g., HCG beta subunit-based monitoring);
* All subjects and their partners voluntarily use contraception as deemed effective by the investigator for at least 90 days from the first dose of the investigational drug to the last dose of the investigational drug (Appendix I); no sperm or egg donation is planned by the subject for at least 6 months from the screening period to the last dose of the investigational drug.
* Subjects can understand the informed consent form, volunteer to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Subjects have had severe allergic reaction related to the investigational drug during the TLL-018-301 study;
* Subjects have had herpes zoster, a major cardiovascular event (MACE), thromboembolism, or lymphoproliferative disorders from the time of TLL-018-301 study to the screening of OLE study;
* Subjects have a clinically significant cardiovascular, respiratory, or any other serious and/or non-stable disease, and there is security risk for subjects to participate in this study judged by the investigator;
* Subjects have abnormal and clinically significant laboratory test values at screening;
* Subjects who have taken traditional Chinese medicines, csDMARDs, immunosuppressive drugs, potent opioids, and other JAK inhibitors (except the investigational drugs in TLL-018-301 study) within 1 week before taking the first dose of the investigational drug in OLE study;
* Subjects have treated with flunomide, any bDMARDs, interferon, and other injected immunosuppressive drugs from TLL-018-301 study to the screening of OLE study;
* Subjects who have received any live vaccine within 2 months prior to taking the first dose of the investigational drug or who plan to receive a live vaccine during the study;
* Subjects have had active tuberculosis infection without evidence of clinical cure; have suspected tuberculosis symptoms judged by the investigator; have latent tuberculosis infection (LTBI) but not received preventive treatment regimens within 3 years prior to screening or not completed a course of therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of occurrences and Percentage of Participants with AEs and SAEs | At Weeks 6, 12, 24, 36, 48, 60, 72, 78
  Evaluation includes vital signs, physical examination, ECG examination, laboratory tests, AE, SAE, etc.

SECONDARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response Over Time | At Weeks 12, 24, 36, 48, 60, 72, 78
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  >=50% improvement in 68-tender joint count; >=50% improvement in 66-swollen joint count; >=50% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity Patient global assessment of disease activity Patient assessment of pain Health Assessment Questionnaire - Disability Index (HAQ-DI) High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response Over Time | At Weeks 12, 24, 36, 48, 60, 72, 78
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  >=20% improvement in 68-tender joint count; >=20% improvement in 66-swollen joint count; >=20% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity Patient global assessment of disease activity Patient assessment of pain Health Assessment Questionnaire - Disability Index (HAQ-DI) High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response Over Time | At Weeks 12, 24, 36, 48, 60, 72, 78
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  >=70% improvement in 68-tender joint count; >=70% improvement in 66-swollen joint count; >=70% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity Patient global assessment of disease activity Patient assessment of pain Health Assessment Questionnaire - Disability Index (HAQ-DI) High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants Achieving Low Disease Activity (LDA) Based on Disease Activity Score-28 (DAS28[CRP]) Over Time | At Weeks 12, 24, 36, 48, 60, 72, 78
  Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28) + 0.36*natural log(hsCRP+1) + 0.014*participant's global assessment of disease activity + 0.96. Scores ranged 0-9.4, where lower scores indicated less disease activity.
Percentage of Participants Achieving Clinical Remission (CR) Based on Disease Activity Score-28 (DAS28[CRP]) Over Time | At Weeks 12, 24, 36, 48, 60, 72, 78
  The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (measured on a VAS from 0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 (CRP) range from 0 to approximately 10, where higher scores indicate more disease activity.
  Clinical remission is defined as a DAS28(CRP) score < 2.6.
Change From Baseline in Disease Activity Score Based on CRP (DAS28 [CRP]) Over Time | Baseline (of the preceding TLL-018-301 study）and Weeks 12, 24, 36, 48, 60, 72, 78
  The disease activity score-28-CRP (DAS28 [CRP]) assesses RA disease activity based on a continuous scale of combined measures of 28 tender joint counts (TJC28), 28 swollen joint counts (SJC28), C-reactive protein (CRP), and the patient global assessment of disease activity (measured on a visual analog scale from 0 to 100 mm). DAS28(CRP) scores range from 0 to approximately 10 where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Over Time | Baseline (of the preceding TLL-018-301 study）and Weeks 12, 24, 36, 48, 60, 72, 78
  The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
Change From Baseline in Clinical Disease Activity Index (CDAI) Over Time | Baseline (of the preceding TLL-018-301 study）and Weeks 12, 24, 36, 48, 60, 72, 78
  The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, and Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. A negative change from Baseline indicates improvement in disease activity.
Change From Baseline in Simplified Disease Activity Index (SDAI) Over Time | Baseline (of the preceding TLL-018-301 study）and Weeks 12, 24, 36, 48, 60, 72, 78
  The simplified disease activity index (SDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm and hsCRP (mg/dL). The total SDAI score ranges from 0 to 86 with higher scores indicating higher disease activity. A negative change from Baseline indicates improvement in disease activity.
Change From Baseline in Patient's Assessment of Pain Over Time | Baseline (of the preceding 301 study）and Weeks 12, 24, 36, 48, 60, 72, 78
  Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain."
Change From Baseline in Patient's Global Assessment of Disease Activity (PtGA) Over Time | Baseline (of the preceding TLL-018-301 study）and Weeks 12, 24, 36, 48, 60, 72, 78
  The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity.
Change From Baseline in Physician's Global Assessment of Disease Activity (PGA) Changes From Baseline in SF-36 Score | Baseline (of the preceding TLL-018-301 study）and Weeks 12, 24, 36, 48, 60, 72, 78
  The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a visual analog scale (VAS) from 0 to 100 mm, where 0 mm indicates no disease activity and 100 mm indicates severe disease activity.
Changes From Baseline in SF-36 Score Over Time | Baseline (of the preceding TLL-018-301 study）and Weeks 24, 48, 78
  SF-36 score was an evaluation of the functional status for a participant,taping eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Coded numeric values are recoded per the scoring key. All items are scored so that a high score defines a more favorable health state. Each item is scored on a o to 100 range. Items in the same scale are averaged together to create the 8 scale scores.
Changes From Baseline in Morning Stiffness Over Time | Baseline (of the preceding TLL-018-301 study）and Weeks 24, 48, 78
  The VAS is a 100 mm line ranging from 0 mm (no morning stiffness) on the left end and 100 mm (worst morning stiffness) on the right end. Subjects marked on the line to indicate their pain severity. The distance in mm was measured from the left end to the subject's marking. Duration of morning stiffness will be from wake-up time to time of resolution of morning stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No